CLINICAL TRIAL: NCT01519245
Title: Topical Application of Tranexamic Acid to Reduce Post-operative Bleeding in Coronary Artery Bypass Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatoon Health Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 67452-01
Record Dates: First submitted 2012-01-17; First posted 2012-01-26 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery bypass grafting; tranexamic acid; antifibrinolytic; administration, topical; operative blood salvage
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trial Drug (Experimental): Solution containing 2 grams tranexamic acid + normal saline
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Tranexamic Acid — Solution containing 2 grams (20mL) tranexamic acid + normal saline (50mL), for a total volume of 70mL poured over the heart as a 'cardiac bath' prior to sternotomy closure near the end of surgery. Total duration of immersion is approximately 10 minutes, until mediastinal chest tubes are connected to suction.
  Arms: Trial Drug
Drug: normal saline — A total volume of 70mL of normal saline poured over the heart as a 'cardiac bath' prior to sternotomy closure near the end of surgery. Total duration of immersion is approximately 10 minutes, until mediastinal chest tubes are connected to suction. Identical in appearance to the trial drug, and is visually indistinguishable.
  Arms: Placebo

SUMMARY:
The goal of this project is to determine whether the use of tranexamic acid, a clot-promoting drug, applied topically over the heart in coronary artery bypass graft surgery (CABG) will reduce post operative blood loss. The investigators' hypothesis is that the use of a tranexamic acid-containing cardiac bath prior to chest closure will result in a statistically significant reduction in blood loss and transfusion requirements in patients who undergo CABG.

DETAILED DESCRIPTION:
Bleeding is expected during major surgeries. In patients who undergo CABG, the risk for bleeding is increased because of the need for intra-operative anticoagulation, or thinning, of patient blood. This anticoagulation is necessary to reduce the risk of thrombosis potentially precipitated by the cardiopulmonary bypass machine, which pumps blood throughout the body while the surgeon operates on the heart.

Strategies are currently used in the operating room to minimize blood loss and the need for allogenic blood transfusion during and after cardiac surgeries. These strategies include the use of intravenous antifibrinolytic agents, intra-operative red blood cell salvage devices, and topical fibrin sealants. Although the risk of infection from a blood transfusion is very small with modern methods of blood screening, the risk of developing a transfusion reaction is possible and not predictable. Therefore, it is preferred to avoid administering a blood transfusion unless absolutely necessary.

The use of topical antifibrinolytic agents has been explored to further reduce blood loss in cardiac surgery. Several trials have been published in the literature since 1993 evaluating the efficacy of various antifibrinolytic medications applied topically, as a cardiac bath, prior to chest closure in CABG patients to reduce post-operative blood loss and potential need for blood transfusion.

The applicability of the methodology utilized in these studies, however, is limited in the context of the current Canadian practices of cardiac surgery. Considerable differences in the perioperative strategies of these trials are seen, in comparison to current North American practices of cardiac surgery. These trials also compared use of topically applied antifibrinolytic agents, including the lysine analogue tranexamic acid, to a control in the absence of intravenous antifibrinolytic agents. The use of intravenous lysine analogues to reduce peri-operative bleeding has now become a near-standard of care in CABG patients.

Currently, the only available antifibrinolytic agent in Canada is the lysine analogue tranexamic acid. This drug is widely used administered as an intravenous preparation in cardiac surgery because its safety profile and reduction in blood loss and frequency of blood transfusion.

There is presently no published randomized controlled trial evaluating blood loss in CABG patients who have received intravenous tranexamic acid, plus topical tranexamic acid or placebo.

ELIGIBILITY:
Inclusion Criterion:

* Patients scheduled for elective or urgent CABG of two to six vessels

Exclusion Criteria:

Preoperative:

* Hemoglobin of less than 110g/L
* Under 18 years of age
* Body mass less than 75kg
* Presence of an intra-aortic balloon pump
* Emergency surgery, requiring operative intervention within 24 hours of consultation to the cardiac surgery team
* Need for cardiac surgical intervention in addition to planned CABG (with the exception of patent foramen ovale closure)
* Ejection fraction (EF) of less than 50%, as determined by echocardiogram or angiography
* Pulmonary hypertension with pulmonary artery pressures greater than 60mmHg (as estimated by right ventricular systolic pressure (RVSP))
* Presence of infectious endocarditis
* Hepatic failure with impaired liver function, including International Normalized Ratio (INR) greater than 1.5
* Known diagnosed bleeding disorder
* History of heparin induced thrombocytopenia and thrombosis (HITT)
* Renal failure with pre-operative creatinine greater than 200ml/min or oliguria with urine output less than 10ml/hour
* Allergy to tranexamic acid
* Pregnancy

Intraoperative:

* Discovery of infectious endocarditis
* Need for cardiac surgical intervention in addition to planned coronary CABG
* Development of allergic reaction to tranexamic acid following intravenous infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Brose, MD, FRCPC, Principal Investigator — University of Saskatchewan, Department of Medicine, Division of Hematology

REFERENCES:
- [Background] Abrishami A, Chung F, Wong J. Topical application of antifibrinolytic drugs for on-pump cardiac surgery: a systematic review and meta-analysis. Can J Anaesth. 2009 Mar;56(3):202-12. doi: 10.1007/s12630-008-9038-x. Epub 2009 Feb 12. PMID 19247741
- [Background] Abul-Azm A, Abdullah KM. Effect of topical tranexamic acid in open heart surgery. Eur J Anaesthesiol. 2006 May;23(5):380-4. doi: 10.1017/S0265021505001894. Epub 2006 Jan 27. PMID 16438759
- [Background] Baric D, Biocina B, Unic D, Sutlic Z, Rudez I, Vrca VB, Brkic K, Ivkovic M. Topical use of antifibrinolytic agents reduces postoperative bleeding: a double-blind, prospective, randomized study. Eur J Cardiothorac Surg. 2007 Mar;31(3):366-71; discussion 371. doi: 10.1016/j.ejcts.2006.12.003. Epub 2007 Jan 10. PMID 17218108
- [Background] De Bonis M, Cavaliere F, Alessandrini F, Lapenna E, Santarelli F, Moscato U, Schiavello R, Possati GF. Topical use of tranexamic acid in coronary artery bypass operations: a double-blind, prospective, randomized, placebo-controlled study. J Thorac Cardiovasc Surg. 2000 Mar;119(3):575-80. doi: 10.1016/s0022-5223(00)70139-5. PMID 10694619
- [Background] Fawzy H, Elmistekawy E, Bonneau D, Latter D, Errett L. Can local application of Tranexamic acid reduce post-coronary bypass surgery blood loss? A randomized controlled trial. J Cardiothorac Surg. 2009 Jun 18;4:25. doi: 10.1186/1749-8090-4-25. PMID 19538741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients scheduled to undergo elective or urgent CABG at Royal University Hospital between December 1, 2011 and April 30, 2012 were screened for participation. Patients meeting inclusion criteria were approached by a study team member at the time of pre-admission clinic attendance or on the in-patient ward with an invitation to participate.
Pre-assignment Details: Patients meeting inclusion criteria were eligible for study participation. Randomization of consented participants took place by the Clinical Trials Pharmacy on the day of surgery, following confirmation of surgical procedure. The study team could withdraw consented patients prior to randomization and surgery if exclusion criteria were identified.
Groups:
- Trial Drug: Total 70mL solution containing 2 grams tranexamic acid (20mL) + normal saline (50mL)
- Placebo: Normal saline (70mL)
Period: Overall Study
Arm/Group | Trial Drug | Placebo
Started | 24 | 20
Received Pre-pump IV TXA | 21 (Two patients included in in the final analysis did not receive pre-pump IV TXA.) | 18 (All patients meeting inclusion criteria received appropriate dosing, as per protocol.)
Received Post-pump IV TXA | 6 (A break in protocol, dosing was given in the operating room at the surgeon's preference.) | 2 (A break in protocol, dosing was given in the operating room at the surgeon's preference.)
Completed | 23 | 18
Not Completed | 1 | 2
Not completed — Met exclusion criteria, not analysed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trial Drug | Placebo | Total
Number analyzed (Participants) | 23 | 18 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 11 | 26
  >=65 years | 8 | 7 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (8.7) | 62 (10.4) | 62 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 17 | 12 | 29
Region of Enrollment [Number; unit: participants]
  Canada | 23 | 18 | 41
Mass [Mean (Standard Deviation); unit: kilograms] | 92.7 (10.5) | 91.3 (13.2) | 92.2 (11.6)
Height [Mean (Standard Deviation); unit: meters] | 1.7 (0.1) | 1.7 (0.1) | 1.7 (0.1)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (4.2) | 31.2 (5.1) | 31.1 (4.6)
Number of Bypasses [Mean (Standard Deviation); unit: Number of vessels] — Mean number of vessels bypassed per patient.
  Number of vessels | 4.1 (1.0) | 4.3 (1.1) | 4.2 (1.1)
Pre-operative Antiplatelet Use [Number; unit: participants] — Participants receiving Aspirin (ASA) or Plavix (any dose) pre-operatively. Divided in to two categories: discontinuation of antiplatelet agents prior to, or at 7 days before surgery; and more than 7 days before surgery.
  participants
    Off 7 days or less | 22 | 18 | 40
    Off more than 7 days | 1 | 0 | 1
Angina [Number; unit: participants] — Symptomatic angina in weeks leading up to surgery.
  participants
    Yes | 22 | 18 | 40
    No | 1 | 0 | 1
History of Myocardial Infarction [Number; unit: participants] — Diagnosed myocardial infarction at any time in participant's past history.
  participants
    Yes | 9 | 9 | 18
    No | 14 | 9 | 23
Stent in situ [Number; unit: participants] — Any history of participant receiving a coronary vascular stent (bare metal or drug eluding).
  participants
    Yes | 3 | 4 | 7
    No | 20 | 14 | 34
Diabetes [Number; unit: participants] — Diagnosis of Type 1 or 2 diabetes (non-insulin dependent or insulin dependent).
  participants
    Yes | 9 | 7 | 16
    No | 14 | 11 | 25
Dyslipidemia [Number; unit: participants]
  Yes | 17 | 13 | 30
  No | 6 | 5 | 11
Atrial Fibrillation [Number; unit: participants]
  Yes | 0 | 0 | 0
  No | 23 | 18 | 41
Hypertension [Number; unit: participants]
  Yes | 18 | 14 | 32
  No | 5 | 4 | 9
Pre-operative Hemoglobin [Mean (Standard Deviation); unit: g/L] | 147 (13) | 142 (14) | 145 (14)
Pre-operative platelet count [Mean (Standard Deviation); unit: platelets x 10^9/L] | 242 (70) | 234 (62) | 239 (66)
Pre-operative white blood cell (WBC) count [Mean (Standard Deviation); unit: WBC x 10^9/L] | 7.7 (1.9) | 7.9 (3.2) | 7.8 (2.5)
Pre-operative International Normalized Ratio (INR) [Mean (Standard Deviation); unit: International Normalized Ratio] — The ratio of a patient's prothrombin time to a normal (control) sample, raised to the power of the International Sensitivity Index (ISI) value for the analytical system used. The calculated value indicates what a patient's PT ratio would be if it was measured using the primary World Health Organization International Reference reagent. The normal range is 0.8-1.2.
  International Normalized Ratio | 1.0 (0.1) | 1.0 (0.1) | 1.0 (0.1)
Pre-operative Creatinine [Mean (Standard Deviation); unit: umol/L] | 84 (25) | 76 (18) | 81 (23)

OUTCOME MEASURES:

1. Primary Outcome: Total Volume of Blood Loss From Mediastinal Chest Tubes at Time of Removal (Assuming the Total Volume of Loss is Blood).
Description: According to standard practice, research participants were be transferred to the intensive care unit (ICU) for post-operative monitoring. Measurement of chest tube output began immediately on arrival to the ICU. Hourly measurements were recorded. Data collection ended upon chest tube removal, or return to the operating room for exploratory surgery due to massive blood loss. As per ICU protocol, chest tubes were be removed when blood loss was recorded to be less than 200mL after six consecutive hours.
Time Frame: From ICU admission post-operatively to mediastinal chest tube removal (placebo group = 20.6 hours; trial group = 19.8 hours)
Population: A total of 44 consented participants were randomized. Prior to unblinding, 3 of the randomized participants were withdrawn from the study due to discovery of ineligibility criteria (1 EF <50%, 1 weight <75kg, 1 CABG x 7). Therefore, a total 41 patients were included in final analysis.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Trial Drug: Total 70mL solution containing 2 grams tranexamic acid (20mL) + normal saline (50mL)
  Total duration that chest tubes were in-situ before removal = 20 hours (SD 3)
- Placebo: Normal saline (70mL)
  Total duration that chest tubes were in-situ before removal = 21 hours (SD 2)
Arm/Group | Trial Drug | Placebo
Number analyzed (Participants) | 23 | 18
mL | 632 (265) | 789 (216)
Statistical Analysis 1: Comparison: Trial Drug vs Placebo; Intention to Treat principles of data analysis were applied. The two-sided T-test (95% confidence interval) was used for statistical calculation of primary outcomes. The null hypothesis was that no difference in chest tube losses would be found between the topical tranexamic acid and placebo groups in low-risk cardiac patients undergoing CABG; Test type: Superiority or Other; p = 0.0493, t-test, 2 sided

2. Primary Outcome: Number of Units of Packed Red Blood Cells (PRBC) Transfused Following Coronary Artery Bypass Graft Surgery
Description: Research participants were to receive a blood transfusion in the Intensive Care Unit (ICU) post-operatively if hemoglobin reached a nadir of 80g/L, or at the discretion of the intensivist or cardiac surgeon according to patient clinical status. Transfusion was quantified based on the number of units of PRBC received. (1 unit = 1 bag of blood, as prepared by Canadian Blood Services). Clinical status of research participants was followed throughout their duration in the ICU only. Participation in this study ended upon transfer out of the ICU, to the Cardiology Ward.
Time Frame: From ICU admission to transfer to the Cardiology Ward (placebo group = 24.4 hours; trial group = 24.7 hours)
Population: None of the research participants received PRBC transfusion postoperatively in the ICU.
Measure: Number; unit: Unit(s) of PRBC
Arm/Group | Trial Drug | Placebo
Number analyzed (Participants) | 23 | 18
Unit(s) of PRBC | 0 | 0

3. Secondary Outcome: Volume of Blood Loss at 6 Hours
Description: Volume of chest tube loss at 6 hours (assuming the total volume of loss is blood).
Time Frame: 6 hours following admission to the Intensive Care Unit
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Trial Drug | Placebo
Number analyzed (Participants) | 23 | 18
mL | 342 (191) | 417 (163)
Statistical Analysis 1: Comparison: Trial Drug vs Placebo; Intention to Treat principles of data analysis were applied. The two-sided T-test (95% confidence interval) was used for statistical calculation of secondary outcomes. The null hypothesis was that no difference in chest tube losses would be found between the topical tranexamic acid and placebo groups in low-risk cardiac patients undergoing CABG; Test type: Superiority or Other; p = 0.1876, t-test, 2 sided

4. Secondary Outcome: Volume of Blood Loss After 12 Hours
Description: Volume of chest tube loss at 12 hours (assuming the total volume of loss is blood).
Time Frame: 12 hours following admission to the Intensive Care Unit
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Trial Drug | Placebo
Number analyzed (Participants) | 23 | 18
mL | 464 (222) | 570 (157)
Statistical Analysis 1: Comparison: Trial Drug vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0930, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Throughout study period duration, and until last enrolled patient was transferred out of the ICU (December 2, 2011-May 3, 2012).
Description: Development of clinically significant vascular or material thrombosis were considered adverse events (cerebrovascular thrombosis, myocardial infarction, deep venous thrombosis, pulmonary embolism or obstructive clot within the mediastinal chest tubes). No serious or other adverse events were observed throughout the duration of the study period.
Arm/Group | Trial Drug | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/18
Other Adverse Events (participants affected / at risk) | 0/23 | 0/18

LIMITATIONS AND CAVEATS:
* Small sample size
* Low-risk CABG patients enrolled only
* Break in protocol, with pre-pump TXA not given to 2 participants, and post-pump TXA given to 8 participants
* Short study period, with no long-term follow-up data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No